CLINICAL TRIAL: NCT05611684
Title: Nanjing First Hospital, Nanjing Medical University
Brief Title: The Influencing Factors of 12 Week Efficacy of Polyethylene Glycol Losenatide in Type 2 Diabetes Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20220825-03
Record Dates: First submitted 2022-10-23; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-09

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — Aftercare

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polyethylene Glycol Losenatide (Experimental): Trearment for 12 weeks
  Interventions: Drug: Polyethylene Glycol Losenatide

INTERVENTIONS:
Drug: Polyethylene Glycol Losenatide — Treatment 0.2mg QW for 12 weeks
  Other Names: Comparison before and after treatment

SUMMARY:
The effect of polyethylene glycol Losenatide on body fat, insulin resistance, weight, blood sugar, blood lipid, stomach volume and other factors in patients with type 2 diabetes through 12 week follow-up, and explore the factors affecting the efficacy, so as to provide more evidence-based medical basis for drug treatment and benefit patients.

DETAILED DESCRIPTION:
The aim of the study is to investigate the factors influencing the efficacy of 12 week treatment with polyethylene glycol Losenatide in type 2 diabetes patients on the basis of diet and exercise. With the 12 week decrease of HbA1c<0.4% from the baseline as the cut-off value, the patients were divided into HbA1c decrease<0.4% group and HbA1c decrease ≥ 0.4% group. The clinical characteristics, laboratory indicators, blood glucose fluctuation of subgroups and gene spectrum differences between the groups were analyzed to provide reference for clinical accurate drug use.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes was diagnosed according to World Health Organization(WHO) classification or other locally applicable diagnostic criteria.
* At least 8 weeks of simple diet control and physical exercise before screening; Type 2 diabetes patients with stable hypoglycemic drug treatment and insufficient blood glucose control within 8 weeks before screening.
* HbA1c≥7.5%.
* Body mass index (BMI) > 24kg /m2.
* Subjects agreed to maintain scientific diet and exercise habits throughout the study, regularly conduct self blood glucose monitoring (SMBG) and make records.
* Willing to sign the written informed consent and abide by the research protocol.

Exclusion Criteria:

* Any of the following drugs or treatments were used within one year before screening: GLP-1RA, GLP-1 analogues, DPP-4 inhibitors or any other incretin analogues.
* Long term (more than 7 consecutive days) intravenous administration, oral administration and intra-articular administration of corticosteroids received within 2 months prior to visit 1.
* Used drugs with weight control effect or performed surgery that may lead to unstable weight within 2 months before screening, or is currently in the weight loss plan and not in the maintenance stage.
* History of acute and chronic pancreatitis; History of myeloid C-cell carcinoma, MEN 2A or 2B syndrome, or related family history.
* Clinically significant abnormal gastric emptying.
* Any organ system tumors that have been treated or not treated within 5 years prior to visit 1.
* Have received coronary angioplasty, coronary stent implantation, and coronary artery bypass surgery within 6 months prior to visit 1, and have experienced negligent compensatory heart failure (NYHA class III and IV of New York Heart Association), stroke or transient ischemic attack, unstable angina, myocardial infarction, and persistent and clinically significant arrhythmia.
* Acute metabolic complications occurred within 6 months prior to visit 1.
* Before screening, any laboratory test index meets the following standards: glutamic pyruvic transaminase>2.5 times or glutamic oxaloacetic transaminase>2.5 times; eGFR<45ml\/min\/1.73m2； Fasting triglyceride>5.64mmol /L.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
blood sugar changes | 12 weeks
  Effects of polyethylene glycol Losenatide on blood sugar changes in Patients With Type 2 Diabetes Mellitus.
blood lipid changes | 12 weeks
  Efficacy of polyethylene glycol Losenatide on blood lipid changes in patients with type 2 diabetes

SECONDARY OUTCOMES:
Body composition analysis | 12 weeks
  Efficacy of polyethylene glycol Losenatide on body composition changes in patients with type 2 diabetes
Inflammation factors | 12 weeks
  Effects of polyethylene glycol Losenatide on inflammation factors in Patients With Type 2 Diabetes Mellitus,after being intervened for 12 weeks,changes of Inflammation factors were observed, including adiponectin,leptin,IL-1,IL-6,IL-18,TNF-α,ghrelin,asprosin.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, Doctor, Study Director — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Jianhua Ma, Nanjing, Jiangsu, China